CLINICAL TRIAL: NCT04231929
Title: BioPearl™ Microspheres Loaded With Doxorubicin to Treat Patients With Unresectable HCC: Prospective, Single Arm, Multi-centre Post-market Follow-up Study.
Brief Title: BioPearl™ Microspheres Loaded With Doxorubicin: Prospective, Single Arm, Multi-centre Post-market Follow-up Study.
Acronym: BIOPEARL-FIRST
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study cancelled by Sponsor decision
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: T135E5
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; Unresectable; BioPearl®; TACE; Chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Chemoembolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BioPearl™ loaded with doxorubicin (Experimental): Chemoembolization with doxorubicin-loaded BioPearl™ microspheres
  Interventions: Device: Chemoembolization

INTERVENTIONS:
Device: Chemoembolization — First, an angiography of the celiac trunk, superior mesenteric artery and hepatic artery will be obtained by using a peripheral arterial approach.
  Arterial embolization will be performed through catheterization of intrahepatic arteries, as selectively as possible (tumor feeders, subsegmental, segmental). The size of the microcatheter must be consistent with the size of BioPearl™ microspheres used. Microspheres of 200 µm will be be used. They will be loaded with the appropriate dose of doxorubicin injectable solution, mixed with the contrast media and distributed according to the location of the HCC lesions. The endpoint of the procedure will be achieved end when stasis of the feeders is achieved.
  Other Names: TACE

SUMMARY:
The primary objective of the study is to confirm safety and efficacy of BioPearl™ microspheres loaded with doxorubicin in the treatment of patients with unresectable hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
This is a prospective, single arm, multi-centre, post-market study to further assess safety and efficacy in 20 unresectable HCC patients treated with Doxorubicin loaded BioPearl™ microspheres.

After the treatment procedure, all patients will undergo clinical follow-up until disease progression and/or next treatment option after which patients will be followed for survival. Patients will be followed up to a maximum of 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years old.
2. Patient with HCC confirmed by histology or according to the latest applicable version of the EASL criteria.
3. Patient with a single nodular tumor 6 cm or less in longest diameter or patient with no more than three tumor nodules, each 4 cm or less in longest diameter. Infiltrative disease is excluded.
4. BCLC B patient or BCLC A patient not a candidate for curative treatment at the time of study inclusion or who has failed/recurred after resection/ablation.
5. Patient deemed treatable in one session for initial treatment.
6. Normal liver or compensated cirrhosis with preserved liver function (Child-Pugh Class A).
7. Total bilirubin ≤ 2.0 mg/dl.
8. Patient with no ascites or with medically controlled ascites.
9. Adequate renal function (serum creatinine < 1.5 X ULN).
10. Patient has provided written informed consent.

Exclusion Criteria:

1. Patient previously treated with any systemic therapy for HCC.
2. Patient previously treated with a loco-regional therapy for HCC. Prior resection/ablation is allowed as per inclusion criteria 4.
3. Eligible for curative treatment at the time of study inclusion.
4. Advanced liver disease: Child-Pugh's B-C class or active gastrointestinal bleeding, encephalopathy.
5. Advanced tumoral disease: BCLC class C or D (vascular invasion - even segmental, extra-hepatic spread or cancer-related symptoms performance status ≥1).
6. Patient with another primary tumor.
7. Patient with history of biliary tree disease or biliary dilatation.
8. Portal vein thrombosis, porto-systemic shunt, hepatofugal blood flow or absent portal blood flow in the liver area to be treated.
9. Contraindication to multiphasic CT and MRI (e.g. allergy to contrast media).
10. Any other contraindication for embolization procedure or doxorubicin treatment.
11. Patient is currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints.

    Note: Trials requiring extended follow-up for products that were investigational, but have become commercially available since then, are not considered investigational trials.
12. In the Investigator's opinion patient has (a) co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study.
13. Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3-4-5 adverse events related with procedure or study device | 4 weeks
  Safety by monitoring and evaluating all grade 3-4-5 adverse events related with procedure or study device
Tumor response | 4 weeks
  Tumor response rate assessed by mRECIST criteria
Tumor response | 12 weeks
  Tumor response rate assessed by mRECIST criteria

SECONDARY OUTCOMES:
Technical success | 1 day
  Ability to reach stasis in the treated tumor feeding arteries during chemoembolization procedure
Time to progression of treated tumor(s) | 3 years
  Time from treatment to progression of the treated lesion according to mRECIST criteria
Time to un-TACEable progression | 3 years
  Time from treatment to un-TACEable progression of the treated lesion according to EASL criteria
Hepatic progression free survival | 3 years
  Time from treatment to progression anywhere in the liver according to mRECIST criteria or death from any cause
Progression free survival | 3 years
  Time from treatment to progression in the liver or outside the liver or death from any cause
Overall survival | 3 years
  Time from treatment until death from any cause
Best overall response | 3 years
  Best response of treated tumor(s) recorded during the course of the study according to mRECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Gontran Verset, MD, Principal Investigator — CUB Hôpital Erasme; Geert Maleux, MD, Principal Investigator — UZ Leuven; Luc Defreyne, MD, Principal Investigator — UZ Gent
Locations (3):
- Belgium (3):
  - CUB Hôpital Erasme, Brussels
  - UZ Gent, Ghent
  - University Hospital Leuven, Leuven